CLINICAL TRIAL: NCT01418508
Title: Effects of Low Protein Diet Supplemented Keto-/Amino Acid in Preventing the Progression of Chronic Kidney Disease(CKD)- ELPD Study
Brief Title: Effects of Low Protein Diet Supplemented Keto-/Amino Acid in Preventing the Progression of Chronic Kidney Disease (CKD)- ELPD Study
Acronym: ELPD-CKD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Xuemei Li, department of nephrology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELPD-CKD
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- low protein diet (No Intervention): Behavioral: low protein diet 0.6g of proteins per kilo of body weight per day
- low protein diet plusα-keto acid (Experimental): 0.6g of proteins per kilo of body weight per day
  Interventions: Behavioral: low protein diet plus α-keto acid
- very low protein diet plus α-keto acid (Experimental): 0.3g of proteins per kilo of body weight per day
  Interventions: Behavioral: very low protein diet plus α-keto acid

INTERVENTIONS:
Behavioral: low protein diet plus α-keto acid — low protein diet plus α-keto acid 0.6g of proteins per kilo of body weight per day, supplemented with α-keto acid tablets
  Arms: low protein diet plusα-keto acid
Behavioral: very low protein diet plus α-keto acid — very low protein diet plus α-keto acid 0.3g of proteins per kilo of body weight per day, supplemented with α-keto acid tablets
  Arms: very low protein diet plus α-keto acid

SUMMARY:
The purpose of this study is to determine whether low protein diet and very low protein diet supplemented keto-/amino acid is effective in preventing the progression of chronic kidney disease (CKD , stage 3b and 4).

DETAILED DESCRIPTION:
Dietary protein restriction represents a basic therapeutic approach in chronic kidney disease(CKD), by reducing the accumulation of nitrogen catabolic substances, and by delaying the progress of CKD and proteinuria, but the effects of the different degree's protein diet on the renal progression remain to be determined.

The aim of this study is to evaluate the efficacy of low protein diet and α-keto acid tablet in retard the progress of CKD. This is a randomized, open-label, prospective study, 120 patients who meet inclusion and exclusion criteria will be randomized into three groups at the ratio of 1:1:1. Group I patients will receive low protein diet(0.6g/kg BW), group II will receive low protein diet supplemented with α-keto acid, while group III will take very low protein diet(0.3g/kg BW) supplemented with α-keto acid. The changes of glomerular filtration rate in CKD will be evaluated after 1 year treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease in stage 3b and 4(15ml/min/1.73m2<GFR<45 ml/min/1.73m2, estimated by EPI formula) receiving conservative treatment for CKD

Exclusion Criteria:

* With diagnosis of diabetic mellitus;
* Incapable of following study requirements to control diet;
* Glomerular filtration rate < 15 ml/min/1.73m2;
* Hypercalcemia or hyperkalemia (> normal upper limit);
* Other serious disease(eg.heart,lung,brain) within the last 3 months;
* Cardiac failure stage IV NYHA;
* With cirrhosis of liver or obvious symptoms of liver diseases, ALT or AST two times normal upper limit;
* Severe edema or serous cavity effusion;
* Drug abuse;
* Final diagnosis of malignant tumor;
* Receiving the long-term systematic steroid hormone or immunosuppressive agents(eg. Cyclophosphamidum,Cyclosporine, Prograf,Azathioprine) treatment;
* Gestation already, prepares to be pregnant in the period of the trial, lactating women;
* Participate in other product clinical trial within 30 days prior to this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
changes in glomerular filtration rate | 1 year

SECONDARY OUTCOMES:
Compliance to diet | 1 year
Quality of life | 1 year
Cardiovascular morbidity | 1 year
  Cardiovascular morbidity, defined by angina, heart failure, myocardial infarction, left ventricular mass, stroke, blood pressure, lipid profile, calcium/phosphorus/parathormone status and Charlson comorbidity index, at the start of dialysis
Nutritional status | 1 year
  Nutritional status, defined by anthropo-plicometry, biochemistry, body bioimpedance analysis (BIA), subjective global nutritional assessment (SGA), at the start and during the 1st year of dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Xuemei Li, M.D.& Ph.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Hahn D, Hodson EM, Fouque D. Low protein diets for non-diabetic adults with chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 29;10(10):CD001892. doi: 10.1002/14651858.CD001892.pub5. PMID 33118160